CLINICAL TRIAL: NCT03686670
Title: Acceptability Study SMARTphone to Collect Clinical Data Using the Memind App by Patients and Medical Satff.
Brief Title: Acceptability Study by Patients Admitted for Suicide and by Medical Staff for Clinical Data Collection Through an E-health Platform
Acronym: MeMind
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: Memind
Record Dates: First submitted 2018-09-20; First posted 2018-09-27 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2016-08

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study goal is to determine the feasbility and interest of monitoring mental health and non mental health related simptoms in Outpatients in order to prevent suicide.

DETAILED DESCRIPTION:
Taking into account the strengths and pitfalls of existing suicide risk assessment methods, we have designed a system capable to combine EMA and continuous monitoring of patients using the smartphone's and/or wearable's sensors and data entry in order to monitor and predict suicide risk. For example, both poor sleep quality and disturbed appetite are clinical markers of depression, with a bidirectional relationship. Their changes could precede the increase of suicidal behavior as sleep and appetite are both influenced by mood state and regulated by the serotonergic system. Our hypothesis is that tracking mental health simptoms regularly through self-report could serve as a consistent and non-biased shortcut to assess mood state, its biological underpinnings and could potentially predict suicidal behavior.

ELIGIBILITY:
To be eligible for the study, patients must be 18 years or older, attend an outpatient clinic or emergency departments of participating clinical services and owning an android or IOS smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After agreeing to participate, clinician will collect the non-opposition for each patient. Patient with a current suicidal behavior disorder (according to DSM-5), i.e. having attempted suicide in the current year, will be test the application.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of this intensive data capture technology in patients in real world without economical incentives. | 2 month
  acceptability assessed by the AES scale

CONTACTS AND LOCATIONS:
Overall Officials: Sofian BERROUIGUET, Study Director — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No